CLINICAL TRIAL: NCT03327558
Title: Full-replicate Study of APRISO 375 mg Extended-release Capsules Versus the Approved APRISO 375 mg Extended-release Capsules in Healthy Male and Female Subjects
Brief Title: Randomized,Study of APRISO 375 mg Versus the Approved APRISO 375 mg Capsules in Healthy Male and Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VLU-P6-774
Record Dates: First submitted 2017-10-26; First posted 2017-10-31 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

STUDY DESIGN:
Intervention Model Description: Single center, laboratory-blinded, randomized, two-treatment, two-sequence, four-period, full replicate, crossover bioequivalence study
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Apriso 0.375G ER CAP (Experimental): Apriso 0.375G ER Cap
  Interventions: Drug: Apriso 0.375G ER CAP
- APRISO 375 mg extended-release capsules (Active Comparator): APRISO 375 mg ER cap
  Interventions: Drug: APRISO 375 mg extended-release capsules

INTERVENTIONS:
Drug: Apriso 0.375G ER CAP — ER capsule
  Arms: Apriso 0.375G ER CAP
Drug: APRISO 375 mg extended-release capsules — 375 mg extended-release capsules
  Arms: APRISO 375 mg extended-release capsules

SUMMARY:
The objective of this study is to evaluate and compare the bioavailability of mesalamine

DETAILED DESCRIPTION:
The objective of this study is to evaluate and compare the bioavailability of mesalamine and therefore to assess the bioequivalence of 375 mg APRISOTM extended-release capsule manufactured at a new site versus the approved 375 mg APRISOTM extended-release capsule after a single oral dose administration under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female, at least 18 years of age
* Body mass index (BMI) between18.5 and below 32.0 kg/m2 (inclusive)
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, ECG and laboratory tests

Exclusion Criteria:

* Any contraindication to mesalamine according to the applicable labeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Cmax (Maximum observed plasma concentration) | 3 hours after oral dose is taken
  Maximum observed plasma concentration levels used for descriptive analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Valeant Site 01, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided